CLINICAL TRIAL: NCT04138225
Title: Assessing the Ecological Role of Yeasts in the Human Gut and Their Impact on Gastrointestinal Disorders
Brief Title: The Ecological Role of Yeasts in the Human Gut
Acronym: YIG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grace Ward (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Royal Berkshire Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Grace Ward, PhD Researcher, University of Reading
Organization: University of Reading (Other)
Other Study IDs: YIGV1
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Irritable Bowel Syndrome; Inflammatory Bowel Diseases; Gastrointestinal Disease
Keywords: yeast; mycology; gut; microbiota; gastrointestinal disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Healthy participants are those without IBS, IBD or any other gastrointestinal disorder
- Irritable bowel syndrome (IBS): Participants with Rome IV diagnosed IBS
- Inflammatory bowel disease (IBD): Patients with IBD - either ulcerative colitis (UC) or Crohn's disease (CD)

SUMMARY:
Irritable bowel syndrome (IBS) and inflammatory bowel disease (IBD) (categorised into Crohn's disease (CD) and ulcerative colitis (UC)) are chronic gut disorders with debilitating symptoms that profoundly impact quality of life, healthcare systems and the economy through lost work days. IBS is common with a prevalence of up to 22%, whereas IBD has a prevalence of 0.3% for CD and 0.5% for UC in Europe. Despite a suggested immunological and genetic aspect of IBD, the causes of IBS and IBD are unknown, however, both have been linked to yeasts in the gut.

Due to their lower abundance (constituting only around 0.1% of the total microorganisms in the gut) yeasts have been less studied than bacteria. More recently, significantly altered diversity and composition of yeasts have been identified in IBS and IBD but further investigation is required to fully develop the role of yeasts in the gut.

This observational study will assess yeasts and their function in the gut, comparing diseased subjects with healthy controls. The overall aim is to determine if yeasts could be targeted as a potential therapeutic for IBS and IBD to provide relief to sufferers as well as reducing the burden on healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-60 years old.
* Either healthy or diagnosed with a gut disorder: Irritable Bowel Syndrome (IBS) or Inflammatory Bowel Disease (IBD) which may include Crohn's disease or ulcerative colitis.
* In good general health.
* Provided written informed consent and willing to participate in this study.

Exclusion Criteria:

* Received antibiotics in the previous six months.
* Consume prebiotics or probiotics on a regular basis (at least 3 times per week) in the last 2 weeks or intend to throughout the course of the study. (Examples of these include: Multibionta multivitamins, Danone Actimel yoghurt drink; Danone Activia yoghurt; Yakult fermented milk drink; Kellogg's Rice Krispies multigrain and Muller Vitality yoghurts/drinks).
* Current use of immunosuppressive drugs.
* Use of other medication which affects gastrointestinal motility and/or gut discomfort.
* History of alcohol or drug misuse.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University, community and primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-09-23 (Actual); Primary Completion 2020-05-23 (Estimated); Study Completion 2021-09-23 (Estimated)

PRIMARY OUTCOMES:
Yeast species in gut | Baseline
  Measured from stool samples using fluorescence in situ hybridisation
Metabolic profile | Baseline
  Measures from stool, urine and blood samples using nuclear magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Calprotectin | Baseline
  Measured using ELISA
Lactorferrin | Baseline
  Measured using ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom